CLINICAL TRIAL: NCT05369234
Title: Effects of Oral Aloe Vera Juice on Chemotherapy and Radiation-induced Oral Mucositis and Esophagitis: a Single-blind Randomized Controlled Trial
Brief Title: Effects of Oral Aloe Vera Juice on Chemotherapy and Radiation-induced Oral Mucositis and Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Covenant Health Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-404 INV Aloe_Oncology
Record Dates: First submitted 2022-04-28; First posted 2022-05-11 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Oral Cavity Cancer; Head and Neck Cancers - Tonsils; Esophageal Cancer; Laryngeal Cancer; Oropharynx Cancer; Mediastinal Cancer; Chest Wall Tumor; Radiation Mucositis
MeSH Terms: conditions — Mouth Neoplasms; Esophageal Neoplasms; Laryngeal Neoplasms; Oropharyngeal Neoplasms; Mediastinal Neoplasms | interventions — Salts; Sucralfate

STUDY DESIGN:
Intervention Model Description: Cohort 1-Lip,oral cavity, hard palate, tongue, tonsil, pharyngeal, laryngeal, neck cancers receiving chemotherapy and radiation therapy will be randomized to receiving either aloe vera juice + standard of care treatments or standard of care treatments.
  Cohort 2--Esophageal, mediastinal, chest wall cancers receiving chemotherapy and radiation will be randomized to receiving aloe vera juice + standard of care treatments or standard of care treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1--Arm 1 (Experimental): Aloe Vera Juice + Standard of Care Treatments Swish and spit ¼ cup (2 ounces) of 100% aloe vera juice 3 times per day, 7 days per week as first line treatment, standard of care agents added as needed
  Interventions: Dietary Supplement: 100% Aloe Vera Juice; Combination Product: Magic Mouthwash; Combination Product: Salt and Baking soda rinse; Drug: Carafate
- Cohort 1--Arm 2 (Active Comparator): Standard of Care Treatments Use salt and baking soda rinses, Magic Mouthwash, Carafate, etc.
  Interventions: Combination Product: Magic Mouthwash; Combination Product: Salt and Baking soda rinse; Drug: Carafate
- Cohort 2--Arm 1 (Experimental): Aloe Vera Juice + Standard of Care Treatments Drink ¼ cup (2 ounces) of 100% aloe vera juice 3 times per day, 7 days per week as first line treatment, standard of care agents added as needed
  Interventions: Dietary Supplement: 100% Aloe Vera Juice; Combination Product: Magic Mouthwash; Combination Product: Salt and Baking soda rinse; Drug: Carafate
- Cohort 2-- Arm 2 (Active Comparator): Standard of Care Treatments Use salt and baking soda rinses, Magic Mouthwash, Carafate, etc.
  Interventions: Combination Product: Magic Mouthwash; Combination Product: Salt and Baking soda rinse; Drug: Carafate

INTERVENTIONS:
Dietary Supplement: 100% Aloe Vera Juice — George's 100% Aloe Vera Liquid Supplement
  Arms: Cohort 1--Arm 1; Cohort 2--Arm 1
Combination Product: Magic Mouthwash — Magic Mouthwash
Combination Product: Salt and Baking soda rinse — Mouth rinse made with salt and baking soda
Drug: Carafate — Carafate taken as a slurry

SUMMARY:
As mentioned above, several prior studies have shown the positive effects of oral use of aloe vera juice in managing chemotherapy and radiation-induced oral mucositis and esophagitis. This study aims to add to the existing body of research around aloe vera juice and its effects on oral mucositis and esophagitis. The intention is to determine whether aloe vera juice should be considered as part of standard treatment.

DETAILED DESCRIPTION:
Oral mucositis and esophagitis are side effects of both chemotherapy and radiation that can interfere with a patient's ability to eat, drink, and maintain weight. They can significantly impact quality of life as well as creating the need for treatment breaks. Treatment breaks decrease the efficacy of treatment. A suspected method of treatment is aloe vera juice. Several prior studies have shown the positive effects of oral use of aloe vera juice in managing chemotherapy and radiation-induced oral mucositis and esophagitis. Aloe vera, or aloe barbadensis miller as it is known in the botanical world, is a succulent plant used in traditional medicine.

In this study, the aloe vera juice that will be utilized by the patients is George's 100% Aloe Vera Juice, manufactured by Warren Laboratories. This aloe vera juice has been fractionally distilled to remove anthraquinone and other compounds that can cause nausea, abdominal cramping, and diarrhea, as well as bitter, unpleasant taste.

This study aims to add to the existing body of research around aloe vera juice and its effects on oral mucositis and esophagitis. The intention is to determine whether aloe vera juice, in combination with standard treatments, is more effective in management of oral mucositis and esophagitis than standard treatment alone. If so, aloe vera offers a natural, cost-effective option for managing radiation and chemotherapy side effects.

Patients in arm 1 of cohort 1 or 2 will be given 3 gallons of George's 100% Aloe Vera Liquid Supplement, free of cost, to utilize throughout treatment. Patients in cohort 1, arm 2 will be asked to swish and spit ¼ cup (2 ounces) of the aloe vera juice 3 times per day, 7 days per week while they are on radiation treatment. Patients in cohort 2, arm 2 will be asked to drink ¼ cup (2 ounces) of aloe vera juice 3 times per day, 7 days per week while they are on chemotherapy and radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* must have signed and dated an IRB approved consent form that conforms to federal and institutional guidelines
* Age >/= 18 years
* Confirmed lip, oral cavity, hard palate, tongue, tonsil, pharyngeal, neck, esophageal, mediastinal, and/or chest wall cancers
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Men treated or enrolled on this protocol must agree to use adequate contraception prior to the study, for the duration of study participation.

Exclusion Criteria:

* Patients who are not on concurrent chemotherapy and radiation.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to aloe vera juice.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women or women who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Prevention of Oral Mucositis and Esophagitis | 10 weeks
  to determine whether to add oral aloe vera juice to standard of care treatments for lip, oral cavity, hard palate, tongue, tonsil , pharyngeal, laryngeal, neck , esophageal, mediastinal, and chest wall cancers will help prevent oral mucositis and esophagitis symptoms while patients undergo radiation therapy. Symptoms will be assessed using the CTCAE v. 5.0 weekly while on treatment to determine if the addition of aloe vera juice impacts these symptoms when compared to subjects that don't receive aloe vera juice.
Management of Oral Mucositis and Esophagitis | 10 weeks
  to determine whether to add oral aloe vera juice to standard of care treatments for lip, oral cavity, hard palate, tongue, tonsil , pharyngeal, laryngeal, neck , esophageal, mediastinal, and chest wall cancers will help manage oral mucositis and esophagitis symptoms while patients undergo radiation therapy. Symptoms will be assessed using the CTCAE v. 5.0 weekly while on treatment to determine if the addition of aloe vera juice impacts these symptoms when compared to subjects that don't receive aloe vera juice.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Scaperoth, MD, Principal Investigator — Covenant Health Cancer Center
Locations (1):
- Thompson Cancer Survival Center Radiation Oncology Services, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
The data analysis will be shared upon completion of the study through a medical publication however at this time the exact plan and what documents is unknown.
Supporting Information: CSR